CLINICAL TRIAL: NCT06533449
Title: Development of the Couplet Care Bassinet to Support Safe Implementation of Skin-to-skin Contact and rooming-in on Postnatal Units
Brief Title: Development of the Couplet Care Bassinet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Couplet Care LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00316391; R44HD097017 (NIH)
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Breastfeeding; Sleep; Patient Satisfaction
Keywords: skin-to-skin; rooming-in; breastfeeding; sleep; bassinet; Cesarean Section
MeSH Terms: conditions — Breast Feeding; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The study will enroll 250 mother-infant pairs at the research location (total n=500, 250 mothers and the infants (250). Half of the pairs (n=250; 125 mothers, 125 infants) will be allocated the Couplet Care Bassinet from enrollment on the postnatal unit through discharge. The other half (n=250; 125 mothers, 125 infants) will be enrolled and assessed as controls with the standard bassinet used at the research site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Couplet Care Bassinet (Experimental): 125 mother-infant pairs will be assigned the Couplet Care bassinet. This bassinet has adjustability features to allow for bassinet positioning over the mother to enable access to the baby, secures the tub in the frame, and has a wall with access points.
  Interventions: Device: Couplet Care Bassinet
- Standard Bassinet (Active Comparator): 125 mother-infant pairs will be assigned the current hospital bassinet offered at the research site. The current bassinet is an unanchored acrylic tub with high walls on a wheeled cart with some storage.
  Interventions: Device: Standard Bassinet

INTERVENTIONS:
Device: Couplet Care Bassinet — Couplet Care Bassinet
  Arms: Couplet Care Bassinet
Device: Standard Bassinet — Standard Bassinet
  Arms: Standard Bassinet

SUMMARY:
The goal of this study is to evaluate the impact of the Couplet Care bassinet on maternal-infant outcomes in the postnatal hospital setting.

The main question this study aims to answer is: Does the Couplet Care bassinet have better maternal-infant outcomes compared to the standard bassinet?

The mother participants will:

-be surveyed about experiences with and use of the bassinet including: the mother's sleep, breastfeeding, calls to staff, infant location, and satisfaction.

Charts will be reviewed for additional outcomes.

Hospital staff and administrators will be surveyed about experiences with the bassinet.

DETAILED DESCRIPTION:
The current study is a Phase II evaluation of the Couplet Care bassinet, designed by Couplet Care Limited Liability Corporation (LLC), a novel infant clinical bassinet designed to support safe implementation of skin-to-skin contact and rooming-in on postnatal units. Until recently, the standard of hospital care for healthy term newborns was to be observed and cared for by maternity staff in a nursery with other infants. However, as detailed in the World Health Organization (WHO) / United Nations International Children's Emergency Fund (UNICEF) report Ten Steps for Successful Breastfeeding, it is now recommended that mothers and infants "room-in" together 24 hours per day, with one hour of separation allowable for procedures outside of the postnatal unit room. As a result, the practice of nursery care is no longer recommended nor facilitated. However, most bassinets in United States (U.S.) hospitals are still designed for use by ambulatory nursery staff, rather than by mobility-impaired new mothers. Current bassinets were not designed for patient use and restrict maternal access to the infants and introduce infants to increased risk of physical injury. Bassinet tubs can tip under the weight of mothers' arms and the height of the tub walls can compromise infant handling. Often, new mothers are required to either substantially twist the body to access the infant or get up out of bed to reach the infant, despite being in immediate postpartum period and needing to heal. Such actions can cause new mothers to experience unnecessary frustration, pain, or even injury. This is especially critical to the one-third of U.S. women who deliver by cesarean section, as the mother's limited ability to move and postpartum pain hinder timely and safe infant care, undermine breastfeeding, impede the mother's own recovery, and contribute to risk of infant falls and suffocation. The substantial difficulty maneuvering infants in and out of conventional bassinets, coupled with the pain and fatigue felt by new mothers, increase the risk of 1) infant drops, and 2) falling asleep with infants in unsafe arrangements. To address these gaps in safety Couplet Care has developed a novel bassinet that allows mothers to position infants over the mother's bed and handle the infants independently.

To ensure usability and safety, the Couplet Care bassinet design incorporates (1) a lower tub wall with access points, making it easier for a mother to reach her infant, (2) adjustability features that allow for bassinet positioning over the mother, and (3) a design that secures the tub into the frame.

In this phase of the project, the researchers will build on insights of Phase I to refine Couplet Care bassinet design, so it is manufacturable and compliant with Food and Drug Administration (FDA) regulations. Next, the Study Team component of the study will:

1. Evaluate the impact of the Couplet Care bassinet on maternal-infant patient outcomes in a powered randomized controlled trial (RCT)
2. Evaluate the usability and adoptability of the device from clinician perspectives. Successful accomplishment of this Phase II effort will position the Couplet Care bassinet for commercialization, delivering a bassinet that promotes safe mother-infant connection during rooming-in, while reducing the risk of infant drops/falls and suffocation, maternal waking from unmet infant needs, and demands on nurses for assistance for non-medical needs.

ELIGIBILITY:
Inclusion Criteria: (from protocol)

* postpartum female participant
* at least 18 years of age
* who can communicate in English

Exclusion Criteria:

* If postpartum female has had multiple infants (twins or more) or
* participant has an infant who is not rooming-in, such as for infant or maternal intensive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women giving birth
Enrollment: 500 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maternal reported infant wakings | Up to 3 days (until discharge)
  Number of times mothers report infant waking

SECONDARY OUTCOMES:
Post-Partum pain levels | Up to 3 days (until discharge)
  reported pain level from participants to medical staff on a scale of 1-10. Higher score indicates higher pain.
Infant feeding substance | Up to 3 days (until discharge)
  Type of feeding substance (participant's own milk, donor human milk, formula use, combination)
Length of postpartum hospitalization | Up to 3 days (until discharge)
  Length of hospitalization
Number of minutes infants were outside of the post-natal unit | Up to 3 days (until discharge)
  Number of minutes infants were outside of the post-natal unit (rooming-in)
Breastfeeding frequency | Up to 3 days (until discharge)
  Breastfeeding frequency
Breastfeeding duration (minutes) | Up to 3 days (until discharge)
  Breastfeeding duration
Number of calls to clinical staff | Up to 3 days (until discharge)
  number of calls by study participants to clinical staff

OTHER OUTCOMES:
Clinician usability assessment | 1 year
  Clinician usability assessment table; clinician must rate 13 statements regarding usability of the bassinet on a scale of 1 to 5 in which 1 is "strongly disagree" and 5 is "strongly agree." Score range 13-65; higher score higher usability
Administrator adoptability assessment | 1 year
  Adoptability table in which administrators rate 4 statements regarding adoptability of the bassinet on a scale of 1 to 5 with 1 being "strongly disagree" and 5 being "strongly agree." Score range 4-20,higher score higher adoptability.
Satisfaction with Bassinet Design | 1 year
  Participants, clinicians, and administrators will be provided open ended questionnaires regarding the design of the bassinet and satisfaction with bassinet use. The participants will be asked two questions to rate the bassinet on ease of use and design on a scale of 1 to 10 with 1 being "not at all" and 10 being "very much". Score range 2-20.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Tomori, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tully KP, Ball HL. Postnatal unit bassinet types when rooming-in after cesarean birth: implications for breastfeeding and infant safety. J Hum Lact. 2012 Nov;28(4):495-505. doi: 10.1177/0890334412452932. Epub 2012 Aug 22. PMID 22914755
- [Background] Tully KP, Ball HL. Maternal accounts of their breast-feeding intent and early challenges after caesarean childbirth. Midwifery. 2014 Jun;30(6):712-9. doi: 10.1016/j.midw.2013.10.014. Epub 2013 Oct 26. PMID 24252711
- [Background] Taylor, Catherine & Tully, Kristin & Ball, Helen. (2015). Night-time on a postnatal ward: experiences of mothers, infants, and staff.
- [Background] Seashore C, Tully KP. Preventing Newborn Falls and Improving Care for Postpartum Women and Their Newborns. Hosp Pediatr. 2018 Sep;8(9):593-594. doi: 10.1542/hpeds.2018-0121. Epub 2018 Aug 1. No abstract available. PMID 30068525
- [Background] Grant D. The "Quiet Revolution" and the cesarean section in the United States. Econ Hum Biol. 2022 Dec;47:101192. doi: 10.1016/j.ehb.2022.101192. Epub 2022 Oct 17. PMID 36351359
- [Background] Brooke J. SUS-A quick and dirty usability scale. Usability evaluation in industry 1996;189(194):4-7
- [Background] Crenshaw JT. Healthy Birth Practice #6: Keep Mother and Baby Together- It's Best for Mother, Baby, and Breastfeeding. J Perinat Educ. 2014 Fall;23(4):211-7. doi: 10.1891/1058-1243.23.4.211. PMID 25411542
- [Background] Consales A, Crippa BL, Cerasani J, Morniroli D, Damonte M, Bettinelli ME, Consonni D, Colombo L, Zanotta L, Bezze E, Sannino P, Mosca F, Plevani L, Gianni ML. Overcoming Rooming-In Barriers: A Survey on Mothers' Perspectives. Front Pediatr. 2020 Feb 21;8:53. doi: 10.3389/fped.2020.00053. eCollection 2020. PMID 32154198
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Background] McKeever J, Fleur RS. Overcoming barriers to Baby-Friendly status: one hospital's experience. J Hum Lact. 2012 Aug;28(3):312-4. doi: 10.1177/0890334412440627. Epub 2012 May 17. PMID 22596059
- See also: WHO/UNICEF Statement — https://iris.who.int/bitstream/handle/10665/39679/9241561300.pdf?sequence=1&isAllowed=y